CLINICAL TRIAL: NCT05438654
Title: Improvement of Diagnostic Approach Using PoCUS for Right Upper Quadrant Abdominal Pain Management in the Emergency Department: A Prospective Study
Brief Title: Improvement of Diagnostic Approach Using PoCUS for Right Upper Quadrant Abdominal Pain
Acronym: DARUQUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DARUQUS
Record Dates: First submitted 2022-06-13; First posted 2022-06-30 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Abdominal Pain
Keywords: Point of Care Ultrasound; Right upper quadrant abdominal pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Intervention Model Description: One group of patients suffering from right upper quadrant abdominal pain will undergo the intervention (Point of care ultrasound of the right upper quadrant). Diagnostic approach will be registered on a case report form (part 1 and part 2) before and after the intervention on a patient. In light of final diagnosis, an adjudication committee will then evaluate the best diagnostic approach, blind to intervention for each patient.
Masking Description: In light of final diagnosis, an adjudication committee will evaluate the best diagnostic approach, blind to intervention for each patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort of patients presenting to emergency department with abdominal right upper quadrant pain (Other): This study is a single arm study analyzing a prospective population of patients presenting at the emergency department complaining of non-traumatic right upper quadrant abdominal pain. The analysis of the diagnostic approach will take place before and after the intervention on a same patient. The intervention is the use of Point of Care Ultrasound bedside.
  Interventions: Diagnostic Test: Point of care ultrasound

INTERVENTIONS:
Diagnostic Test: Point of care ultrasound — Abdominal PoCUS use according to the following protocol:
  PoCUS assessment of the right lung base PoCUS assessment of Morrison's pouch PoCUS assessment of gallbladder PoCUS assessment of right kidney (comparison to left kidney acceptable) PoCUS assessment of small bowel

SUMMARY:
Many medical specialties and paramedical fields are increasingly using point-of-care ultrasound (PoCUS). In daily practice, abdominal pain accounts for 7% to 10% of emergency department consultations, while the mean reported prevalence of abdominal pain in family physician consultations is 2.8%. PoCUS can be used in a variety of ways during abdominal physical examinations, and most scientific societies encourage its use to address a specific clinical question rather than provide a diagnosis, which is usually confirmed by comprehensive ultrasound in radiology. The integration of PoCUS into clinical examination raises the issue of PoCUS accuracy to improve the diagnostic approach as opposed to PoCUS diagnostic accuracy itself. Considering the wide range of differential diagnoses associated with right upper quadrant pain, this multicenter prospective study protocol aims to evaluate the improvement of the diagnostic approach using PoCUS in patients presenting at an emergency department with right upper quadrant abdominal pain. In light of the final diagnosis at 1-month follow-up, two members of an adjudication committee will blindly choose between two case report forms: one filled in before PoCUS and the other completed after the use of PoCUS by the investigator in charge of a patient suffering from right upper quadrant abdominal pain. The hypothesis that PoCUS enhances diagnostic approaches by 18% will be reached if 74.8% of the better diagnostic approaches are in favor of the case report form filled in after PoCUS.

DETAILED DESCRIPTION:
1. Background Many medical specialties and paramedical fields are increasingly using point-of-care ultrasound (PoCUS). PoCUS is a pillar of clinical evaluation along with inspection, palpation, percussion, and auscultation, and it has become essential in daily clinical practice, as it enhances differential diagnosis. In a position statement published in 2015, the American Academy of Emergency Medicine followed by the European Federation of Societies for Ultrasound in Medicine and Biology in 2016 recommended the inclusion of PoCUS in the curricula of medical schools to improve the learning of core concepts and enhance students' understanding of physical examinations. The integration of PoCUS into clinical examination raises the issue of PoCUS accuracy to improve the diagnostic approach as opposed to the issue of PoCUS diagnostic accuracy itself.

   In daily practice, abdominal pain accounts for 7% to 10% of emergency department consultations, while the mean reported prevalence of abdominal pain in family physician consultations is 2.8% according to a recent systematic review. PoCUS can be used in many ways during abdominal physical examinations, and most scientific societies encourage its use to address a specific clinical question rather than to provide a diagnosis, which is usually confirmed by a comprehensive ultrasound in radiology. For this reason, it is necessary to evaluate PoCUS accuracy in order to improve the diagnostic approach.

   Among abdominal pain, right upper quadrant pain evokes a large differential diagnosis. PoCUS is a valuable tool to investigate right upper quadrant abdominal pain, as it can orientate the investigator toward the presence of free fluid, lung involvement, aortic aneurysm, gallbladder involvement, hydronephrosis, or small bowel obstruction.

   The primary objective of this study is to evaluate the contribution of PoCUS to the clinical examination of patients presenting in an emergency department with right upper quadrant abdominal pain. The secondary outcomes are the influence of PoCUS on the choice and number of additional complementary diagnostic examinations, its influence on the physicians' coefficient of certainty in terms of the diagnostic approach, differential diagnosis, and initiated treatment, and finally, the influence of patients' characteristics or PoCUS findings on the primary outcome.
2. Method

   1. Trial design This study is an interventional multicenter prospective study assessing the improvement of the diagnostic approach using PoCUS as part of the clinical examination for patients presenting in an emergency department with right upper quadrant abdominal pain.

      The interventional nature of the study is motivated by the lack of clear guidelines in Belgium regarding the integration of PoCUS into the standard of care contrary to other countries in Europe and North America.

      Follow-up at 1 month based on patients' medical files and telephone interviews (patient and/or treating physician) is required to determine the final diagnosis.

      The study will take place in two tertiary university centers (Cliniques Universitaires Saint Luc, Bruxelles and Centre hospitalier universitaire, Liège) as well as three secondary-level hospitals (Hôpital Jolimont Lobbes, Haine Saint Paul; Grand Hôpital de Charleroi, Charleroi; Cliniques Saint-Pierre, Ottignies).
   2. Study procedure Eligibility Patient eligibility will be determined by nurses at triage.

      Any patient presenting with abdominal pain will be evaluated according to the following three questions:
      * Can you show me with your hand where is the pain located?
      * Have you been in pain for less than 11 days?
      * Did you undergo any complementary medical examinations to evaluate the pain before coming to our emergency department (urine sample, blood sample, medical imaging)? Inclusion process Without interfering with the patient triage, the study investigator will assess the patient's eligibility, explain the study, and obtain signed informed consent. The investigator will then verify the inclusion and exclusion criteria and initiate the study process by taking charge of the patient and performing an anamnesis and clinical examination.

      The investigator will fill in the first part of the CRF (Part 1) and place it in a first sealed envelope.

      Intervention process The investigator uses PoCUS according to intervention protocol. The investigator will fill in the second part of the CRF (Part 2) and place it in a second sealed envelope.

      The investigator is not required to limit the PoCUS examination to the PoCUS protocol if the patient's care requires further PoCUS examinations. However, the rest of the PoCUS examination will be performed after the three sections of the CRF are completed and sealed.

      Evaluation process The first adjudication committee will determine the final diagnosis based on the patient's medical file and 1-month follow-up. They have no access to the study data except for question relating to the 1-month follow-up.

      After validating the final diagnosis and anonymizing the data, the second adjudication committee will evaluate the diagnostic approaches. This second adjudication committee is blind to the intervention. Before assessing the diagnostic approach, Parts 1 and 2 of the CRF are anonymized and randomly ordered using the "Randomizer for Clinical Trial Lite" Medsharing, Fontenay-Sous-Bois, France.

      After evaluating the two CRF parts, the members of the second adjudication committee will choose the better diagnostic approach or state that the diagnostic approaches are unchanged.

      After collecting the results, any discrepancies will be adjudicated by a third member according to the same process.

      Study members
      * Investigators The investigators are all emergency physicians who are familiar with PoCUS of the right upper quadrant and who underwent a 2-hour refresher course on the PoCUS process used for this particular study.
      * Adjudication committee members Adjudication committee 1 Three emergency physicians confirm the final diagnoses of patients according to their medical file and 1-month follow-up.

      Adjudication committee 2 Two emergency physicians who are blind to the intervention and independent of the study separately choose the better diagnostic approach based on the CRFs (Part 1, and Part 2). A third member independent of the study may be required to adjudicate any discrepancies after cross-referencing the results.
   3. Sample size A total of 59 patients are needed to show a 18% improvement in the diagnostic approach with a power of 0.9 and an alpha value of 0.05. Considering an attrition rate of 10%, the sample size needed to perform this study is 65 patients. An 18% improvement in the diagnostic process from 56.8% to 74.8% is based on previous publications showing a 56.8% rate of correct diagnosis after anamnesis and clinical examination without PoCUS in non-traumatic abdominal pain and an improvement in the diagnostic accuracy or diagnostic process from 12% to 24% with the use of PoCUS depending on the study.
   4. Statistical method The software IBM SPSS statistics 26.0 (SPSS Inc., Chicago, IL, USA) will be used to analyze the data. Continuous variables describing the study population will be detailed using medians, standard deviations, and minimum and maximum values. Discrete variables will be reported by category as numbers and percentages. The χ² test of independence will be used for comparison between discrete variables. The Wilcoxon-Mann-Whitney test will be used for comparison between continuous variables. The significance level corresponds to a p-value of < 0.05. The 95% confidence intervals will be calculated using the mid-p exact value.

   Primary endpoint will be evaluated using a proportion test performed according to the expected percentage of improvement (18%).
3. Data management

   1. Data collection All the data relating to this study will be collected on paper CRF by the study investigator. Collected data will concern the clinical situation, patient characteristics, test results, and diagnostic approach associated with the coefficients of certainty of the physicians in charge as well as any questions relating to the bedside PoCUS. Any missing data will be collected from the medical file by the inclusion center's principal investigator, coordinating investigator, or research associates.

      Patients will initially be identified on the CRF by their last name, first name, date of birth, file number from the institution where they were included, and an identification number of the study. This identification number will be comprised of a reference for the inclusion center and participant number. After the principal investigators or research associates complete the collection of missing data, patients will henceforth only be identified by their study identification number to anonymize the data.
   2. Data access A list of correspondence between the study identification number and the other identifying data will be kept under the responsibility of the project promoter. This list is kept for the statutory period of time provided for this type of research. The protection of the patients' personal data will be guaranteed by the European General Data Protection Regulation of 27 April 2016 (in application since 25 May 2018), the Belgian Law of 30 July 2018 on privacy protection with regard to the processing of personal data, and the Belgian Law of 22 August 2002 on patient rights.

      A certified good clinical practice will be used with a compliant electronic data management system. The system is connected to the clinical center database management system and protected by the personal identification of authorized users. This distinguishes between users and guarantees data safety.

      Any individual with direct access to the data shall take all the necessary precautions to ensure the confidentiality of the information relating to participants included in the study, particularly with regard to their identity and results. Any individual with direct access to data are subject to professional secrecy. They undertake to never divulge confidential information relating to the study participants and to guarantee the anonymization of the data before transferring it to the database manager and biostatistician. Any data disclosure required by the law or applicable regulations will be done if necessary.
   3. Data storage After completing the data collection and anonymizing the data, they will be added to a file (SPSS 26.0) with access limited by a password. This document will be owned by the project promoter represented by the study coordinator. This person ensures that the documents and data relating to the research are kept for 25 years in accordance with the applicable regulations.
4. Ethics Written documentation explaining the PoCUS procedure and the risks/benefits of undergoing PoCUS will be given to all participants. They will also receive an explanation about data protection.

Ultrasound technology does not put participants at risk during abdominal ultrasound. Indeed, physicians are required to observe the ALARA (as low as reasonably achievable) principle during clinical examinations. Signed written consent to participate in this study will be collected for each participant as recommended by the Additional Protocol to the Convention on Human Rights and Biomedicine Concerning Biomedical Research as well as by the Council of Europe's Steering Committee on Bioethics.

1. Adverse event An adverse event is any untoward medical occurrence including the exacerbation of an existing condition that is not necessarily related to the study itself. Any incidental findings using PoCUS will be reported, and information will be given under medical confidentiality.
2. Insurance Regarding the Belgian law of 7 May 2004, the project promoter will take out insurance to cover any risk incurred by the study's participants

ELIGIBILITY:
Inclusion Criteria:

* > 17 years
* Right upper quadrant abdominal pain < 11 days
* Signed informed consent

Exclusion Criteria:

* Any reason that prevents ultrasound use
* Pregnancy
* Palliative care status or poor prognosis at 1-month follow-up
* Impossibility of 1-month follow-up
* Insufficient knowledge of French or Dutch to understand the informed consent

Secondary exclusion criteria:

* Lost to follow-up
* Previously unknown pregnancy diagnosed during the emergency department consultation
* Emergency of care deemed incompatible with the study process by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Change in diagnostic approach before and after the use of point of care ultrasound | through study completion, at an average of 7 months
  Rate of diagnostic approach considered improved after intervention by the adjudication committee Two independent members of an adjudication committee will evaluate two diagnostic approaches (before and after PoCUS) reported in the case report forms (CRFs) of patients suffering from right upper quadrant abdominal pain in an emergency setting while considering the final diagnosis determined at 1-month follow-up. As the adjudication committee members are blind to the intervention, they do not know which diagnostic approach reported in the CRFs is performed before or after PoCUS.
  For each patient file, the adjudication committee must choose the better diagnostic approach or state that the diagnostic approach is unchanged.

SECONDARY OUTCOMES:
PoCUS influence on the choice of complementary examination(s) | through study completion, at an average of 7 months
  Rate of complementary examination procedure considered to be the most adequate by the adjudication committee blind to the intervention based on the CRFs (before and after PoCUS)
Comparison of the absolute number of complementary examination planned before and after intervention | through study completion, at an average of 7 months
  Comparison of absolute number of complementary examination(s) before and after PoCUS
PoCUS influence on the physicians' coefficient of certainty regarding the diagnostic approach | through study completion, at an average of 7 months
  Percentage of improvement of investigators certainty coefficient for diagnostic approach, measured with a percentage scale (0%-20%-40%-60%-80%-100%), after the intervention PoCUS
PoCUS influence on the physicians' coefficient of certainty regarding the differential diagnosis | through study completion, at an average of 7 months
  Percentage of improvement of investigators certainty coefficient for differential diagnosis, measured with a percentage scale (0%-20%-40%-60%-80%-100%), after the intervention PoCUS
PoCUS influence on the physicians' coefficient of certainty regarding the initiated treatment | through study completion, at an average of 7 months
  Percentage of improvement of investigators certainty coefficient for initiated treatment, measured with a percentage scale (0%-20%-40%-60%-80%-100%), after the intervention PoCUS
PoCUS usefulness qualitatively evaluated by the investigator as:not useful, slightly useful, moderately useful, useful, very useful | through study completion, at an average of 7 months
  percentage of PoCUS in each category - not useful, slightly useful, moderately useful, useful, very useful
Influence of PoCUS findings (hydronephrosis, gallstones, free fluid, aortic aneurysm, small bowel obstruction, pleural effusion, lung interstitial syndrome) on the primary outcome | through study completion, at an average of 7 months
  Rate of diagnostic approach considered improved after intervention by the adjudication committee for each subgroup.
Influence of patients' characteristics (BMI, echogenicity, triage score, pain scale, final diagnosis) on the primary outcome | through study completion, at an average of 7 months
  Rate of diagnostic approach considered improved after intervention by the adjudication committee for each subgroup

CONTACTS AND LOCATIONS:
Overall Officials: Florence Dupriez, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires saint luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meadley B, Olaussen A, Delorenzo A, Roder N, Martin C, St Clair T, Burns A, Stam E, Williams B. Educational standards for training paramedics in ultrasound: a scoping review. BMC Emerg Med. 2017 Jun 17;17(1):18. doi: 10.1186/s12873-017-0131-8. PMID 28623905
- [Background] Totenhofer R, Luck L, Wilkes L. Point of care ultrasound use by Registered Nurses and Nurse Practitioners in clinical practice: An integrative review. Collegian. août 2021;28(4):456-63.
- [Background] Hayward SA, Janssen J. Use of thoracic ultrasound by physiotherapists: a scoping review of the literature. Physiotherapy. 2018 Dec;104(4):367-375. doi: 10.1016/j.physio.2018.01.001. Epub 2018 Feb 2. PMID 29958691
- [Background] Soucy ZP, Mills LD. American Academy of Emergency Medicine Position Statement: Ultrasound Should Be Integrated into Undergraduate Medical Education Curriculum. J Emerg Med. 2015 Jul;49(1):89-90. doi: 10.1016/j.jemermed.2014.12.092. Epub 2015 Apr 29. No abstract available. PMID 25934381
- [Background] Cantisani V, Dietrich CF, Badea R, Dudea S, Prosch H, Cerezo E, Nuernberg D, Serra AL, Sidhu PS, Radzina M, Piscaglia F, Bachmann Nielsen M, Ewertsen C, Saftoiu A, Calliada F, Gilja OH. EFSUMB Statement on Medical Student Education in Ultrasound [long version]. Ultrasound Int Open. 2016 Mar;2(1):E2-7. doi: 10.1055/s-0035-1569413. PMID 27689163
- [Background] Nicholas E, Ly AA, Prince AM, Klawitter PF, Gaskin K, Prince LA. The Current Status of Ultrasound Education in United States Medical Schools. J Ultrasound Med. 2021 Nov;40(11):2459-2465. doi: 10.1002/jum.15633. Epub 2021 Jan 15. PMID 33448471
- [Background] Prosch H, Radzina M, Dietrich CF, Nielsen MB, Baumann S, Ewertsen C, Jenssen C, Kabaalioglu A, Kosiak W, Kratzer W, Lim A, Popescu A, Mitkov V, Schiavone C, Wohlin M, Wustner M, Cantisani V. Ultrasound Curricula of Student Education in Europe: Summary of the Experience. Ultrasound Int Open. 2020 Jun;6(1):E25-E33. doi: 10.1055/a-1183-3009. Epub 2020 Aug 31. PMID 32885138
- [Background] Atkinson P, Bowra J, Lambert M, Lamprecht H, Noble V, Jarman B. International Federation for Emergency Medicine point of care ultrasound curriculum. CJEM. 2015 Mar;17(2):161-70. doi: 10.1017/cem.2015.8. PMID 26052968
- [Background] Cervellin G, Mora R, Ticinesi A, Meschi T, Comelli I, Catena F, Lippi G. Epidemiology and outcomes of acute abdominal pain in a large urban Emergency Department: retrospective analysis of 5,340 cases. Ann Transl Med. 2016 Oct;4(19):362. doi: 10.21037/atm.2016.09.10. PMID 27826565
- [Background] Viniol A, Keunecke C, Biroga T, Stadje R, Dornieden K, Bosner S, Donner-Banzhoff N, Haasenritter J, Becker A. Studies of the symptom abdominal pain--a systematic review and meta-analysis. Fam Pract. 2014 Oct;31(5):517-29. doi: 10.1093/fampra/cmu036. Epub 2014 Jul 1. PMID 24987023
- [Background] Martinez M, Duchenne J, Bobbia X, Brunet S, Fournier P, Miroux P, et al. Deuxième niveau de compétence pour l'échographie clinique en médecine d'urgence. Recommandations de la Société française de médecine d'urgence par consensus formalisé. Ann Fr Médecine D'urgence. juin 2018;8(3):193-202
- [Background] Ma IWY, Arishenkoff S, Wiseman J, Desy J, Ailon J, Martin L, Otremba M, Halman S, Willemot P, Blouw M; Canadian Internal Medicine Ultrasound (CIMUS) Group*. Internal Medicine Point-of-Care Ultrasound Curriculum: Consensus Recommendations from the Canadian Internal Medicine Ultrasound (CIMUS) Group. J Gen Intern Med. 2017 Sep;32(9):1052-1057. doi: 10.1007/s11606-017-4071-5. Epub 2017 May 11. PMID 28497416
- [Background] Smallwood N, Dachsel M. Point-of-care ultrasound (POCUS): unnecessary gadgetry or evidence-based medicine? Clin Med (Lond). 2018 Jun;18(3):219-224. doi: 10.7861/clinmedicine.18-3-219. PMID 29858431
- [Background] Lynch RM. Accuracy of abdominal examination in the diagnosis of non-ruptured abdominal aortic aneurysm. Accid Emerg Nurs. 2004 Apr;12(2):99-107. doi: 10.1016/j.aaen.2003.09.005. PMID 15041011
- [Background] Miller AH, Pepe PE, Brockman CR, Delaney KA. ED ultrasound in hepatobiliary disease. J Emerg Med. 2006 Jan;30(1):69-74. doi: 10.1016/j.jemermed.2005.03.017. PMID 16434339
- [Background] Torres-Macho J, Anton-Santos JM, Garcia-Gutierrez I, de Castro-Garcia M, Gamez-Diez S, de la Torre PG, Latorre-Barcenilla G, Majo-Carbajo Y, Reparaz-Gonzalez JC, de Casasola GG; Working Group of Clinical Ultrasound, Spanish Society of Internal Medicine. Initial accuracy of bedside ultrasound performed by emergency physicians for multiple indications after a short training period. Am J Emerg Med. 2012 Nov;30(9):1943-9. doi: 10.1016/j.ajem.2012.04.015. Epub 2012 Jul 12. PMID 22795427
- [Background] Taylor MR, Lalani N. Adult small bowel obstruction. Acad Emerg Med. 2013 Jun;20(6):528-44. doi: 10.1111/acem.12150. PMID 23758299
- [Background] Ultrasound Guidelines: Emergency, Point-of-Care and Clinical Ultrasound Guidelines in Medicine. Ann Emerg Med. 2017 May;69(5):e27-e54. doi: 10.1016/j.annemergmed.2016.08.457. No abstract available. PMID 28442101
- [Background] membres de la commission des référentiels de la SFMU, Duchenne J, Martinez M, Rothmann C, Claret PG, Desclefs JP, et al. Premier niveau de compétence pour l'échographie clinique en médecine d'urgence. Recommandations de la Société française de médecine d'urgence par consensus formalisé. Ann Fr Médecine Urgence. juill 2016;6(4):284-95
- [Background] Miller DL, Abo A, Abramowicz JS, Bigelow TA, Dalecki D, Dickman E, Donlon J, Harris G, Nomura J. Diagnostic Ultrasound Safety Review for Point-of-Care Ultrasound Practitioners. J Ultrasound Med. 2020 Jun;39(6):1069-1084. doi: 10.1002/jum.15202. Epub 2019 Dec 23. PMID 31868252
- [Background] Booth TC, Jackson A, Wardlaw JM, Taylor SA, Waldman AD. Incidental findings found in "healthy" volunteers during imaging performed for research: current legal and ethical implications. Br J Radiol. 2010 Jun;83(990):456-65. doi: 10.1259/bjr/15877332. Epub 2010 Mar 24. PMID 20335427
- [Derived] Dupriez F, Druez D, Ries A, Stevens F, Penaloza A, Rodrigues de Castro B. Impact of point-of-care ultrasound in right upper quadrant abdominal pain in an emergency department: cost analysis. Acta Clin Belg. 2026 Jan 20:1-9. doi: 10.1080/17843286.2026.2618115. Online ahead of print. PMID 41557443